CLINICAL TRIAL: NCT07087197
Title: A Multicenter, Open-label Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Dosimetry and Efficacy of SKB107 in Subjects With Advanced Solid Tumors With Bone Metastases
Brief Title: A Study of SKB107 in Advanced Solid Tumors With Bone Metastases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SKB107-I-01
Record Dates: First submitted 2025-06-30; First posted 2025-07-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1a：Dose escalation (Experimental): 5 dose levels are tentatively planned for Phase 1a
  Interventions: Drug: SKB107 for injection
- Phase 1b: Dose expansion (Experimental): The dose of SKB107 for injection in Phase 1b is selected based on the Phase 1a monotherapy dose escalation study
  Interventions: Drug: SKB107 for injection

INTERVENTIONS:
Drug: SKB107 for injection — 177Lu-DOTA-IBA is a Radionuclide conjugated drugs (RDC) targeting bone.

SUMMARY:
A multicenter, open-label Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, dosimetry and efficacy of SKB107 in subjects with advanced solid tumors with bone metastases.

DETAILED DESCRIPTION:
This study is a multicenter, open-label Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, dosimetry and efficacy of SKB107 in subjects with advanced solid tumors with bone metastases. The study is divided into two parts: Phase Ia and Phase Ib. The Phase Ia study is the dose escalation phase. The primary objective is to assess the safety and tolerability of a single administration of SKB107 and to determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) based on the occurrence of Dose-Limiting Toxicities (DLTs) associated with SKB107 (if the MTD cannot be determined).The Phase Ib study is the dose expansion phase. The primary objective is to explore the optimal dose, safety, or efficacy of SKB107 at a selected dose level (confirmed as safe by the Safety Review Committee (SRC) and not exceeding the MTD or MAD)

ELIGIBILITY:
Inclusion Criteria:

1. The age should be between 18 years and 75 years at the time of signing the informed consent form (ICF);
2. The Eastern Cooperative Oncology Group (ECOG) performance status score should be ≤ 1;
3. The expected survival period should be ≥ 3 months;
4. Phase Ia: Subjects with advanced solid tumor bone metastases diagnosed by histology or cytology; and the subjects have failed standard treatment, or have no standard treatment, or are intolerant or not applicable to standard treatment;
5. Phase Ib: Subjects with advanced mCRPC diagnosed by histology or cytology;
6. Before the first administration, a 99mTc-MDP bone scan diagnosed multiple bone metastases, and at least one site was confirmed by CT or MRI;
7. Have adequate organ and bone marrow functions;
8. For subjects with reproductive capacity, take effective medical contraceptive measures during the study treatment and within 6 months after the last administration;
9. The subjects voluntarily join this study, sign the informed consent form, and can comply with the visit and related procedures stipulated in the protocol.

Exclusion Criteria:

1. The washout period before the first administration of the study drug was insufficient.
2. Previous received similar radionuclide internal irradiation treatment.
3. Previous received or planned to receive during the study period semi-body external radiotherapy targeting bone metastases.
4. Known "super bone imaging".
5. Known spinal cord compression, or clinical imaging manifestations suggesting impending spinal cord compression.
6. Any cardiovascular or cerebrovascular diseases or cardiovascular risk factors that may affect the treatment of the study drug.
7. Poorly controlled diabetes and hypertension.
8. The toxicity of previous anti-tumor treatment before the first administration has not recovered to ≤ 1 grade (evaluated based on NCI-CTCAE v5.0) or has not reached the level specified in the inclusion/exclusion criteria.
9. Had other malignant tumors within 3 years before the first administration.
10. Subjects with severe and/or uncontrolled concomitant diseases.
11. Active hepatitis B or active hepatitis C.
12. Human immunodeficiency virus (HIV) test positive or having a history of acquired immune deficiency syndrome (AIDS); known active syphilis infection.
13. Subjects with a history of radionuclide/radioactive drug allergy, or allergic to any component of the study formulation.
14. During the screening process before the first administration, the condition deteriorated rapidly, such as significant changes in the investigator's assessment of physical condition, etc.
15. Subjects participating in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an intervention study.
16. Any unstable disease or clinical condition, or any condition that may endanger the safety of the subject or affect the subject's compliance, or any other conditions that the investigator deems inappropriate for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | Up to 3 year

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of SKB107 | Up to 1 week
Dosimetry | Up to 1 week
  To collec the biological distribution of major tissues/organs.
Time to Radiographic Bone Progresion (TTRBP) | Through study completion, an average of 1 year.
  Time from start of treatment to progression of bone lesion (PD) or death, whichever occurs first, during the study period
Radiographic progression-free survival (rPFS) | Through study completion, an average of 1 year
  Time from start of treatment to progression of Disease (PD) or death, whichever occurs first
Overall survival(OS) | Up to 3 years
  Time from start of treatment to death due to any reason
symptomatic skeletal event-free survival (SSE-FS) | Up to 3 years
  Time from start of treatment to the first occurrence of new SSE or death from any cause , whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China